CLINICAL TRIAL: NCT00003298
Title: A Phase II Trial of Neoadjuvant Paclitaxel - Cisplatin Chemotherapy, Surgery and Adjuvant Radiation Therapy and 5-FU/Leucovorin for Gastric Cancer
Brief Title: Chemotherapy, Surgery, and Radiation Therapy in Treating Patients With Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066237; E7296 (Other: Eastern Cooperative Oncology Group); U10CA023318 (NIH); NCT00003298 (Registry Identifier: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2004-01-23 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer
Keywords: stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Platinum; Fluorouracil; Leucovorin; Paclitaxel; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Arm (Experimental): Patients receive 3 courses of preoperative neoadjuvant chemotherapy given on day 1 every 21 days. Courses consist of an intravenous infusion of cisplatin and a 3 hour intravenous infusion of paclitaxel on day 1. Patients then undergo surgery for tumor removal on day 63, followed 4-6 weeks later by one course of daily intravenous bolus leucovorin calcium and fluorouracil for 5 days. Chemotherapy is repeated 4-6 weeks later for the first 4 days of week 1 and the last 3 days of week 5 of radiation therapy given 5 days a week for 5 weeks. Patients receive two more courses, 4 weeks apart, of fluorouracil and leucovorin calcium for 5 days 4-6 weeks after completing radiation treatment.
  Interventions: Drug: cisplatin; Drug: fluorouracil; Drug: leucovorin calcium; Drug: paclitaxel; Procedure: surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Cisplatin was administered as part of the neoadjuvant regimen. It was given at a dose of 75 mg/m² via IV over approximately one hour, on day 1 of each cycle. Three cycles were given.
  Other Names: Platinol; cis-platinum; cisdiamminedichloroplatinum (II); Platinol-AQ; DACP; platinum; CDDP; DDP
Drug: fluorouracil — Postoperative regimen 5-FU, along with Leucovorin, was given by IV bolus, with 5-FU given immediately after the Leucovorin
  Other Names: 5-Fluorouracil; 5-FU; Adrucil; Efudex
Drug: leucovorin calcium — Both 5-FU and Leucovorin will be given via IV bolus, with Leucovorin given immediately before 5-FU.
  Other Names: Leucovorin; Wellcovorin; citrovorum factor; folinic acid; 5-formyl tetrahydrofolate; LV; LCV
Drug: paclitaxel — Paclitaxel was administered as part of the neoadjuvant regimen. It was given at a dose of 175 mg/m² as a 3 hour continuous intravenous infusion on day 1. Three cycles were given.
  Other Names: Taxol®; NSC 125973
Procedure: surgery — The surgical procedure performed involved a radical subtotal or total gastrectomy.
  A complete surgical resection was required
Radiation: radiation therapy — Concomitant chemotherapy and radiation therapy course: 5-FU 400 mg/m²/day + Leucovorin 20 mg/m²/day on days 1-4 of week one and days 1-3 of week 5 of XRT. Combined chemotherapy and radiation therapy were to begin 4 weeks after day 1 of the initial course of chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy, radiation therapy, and surgery may kill more tumor cells. E7296 was conducted to study neoadjuvant chemotherapy and postoperative chemoradiation therapy in patients diagnosed with high-risk gastric cancer using a new neoadjuvant regimen: paclitaxel plus cisplatin. It was hypothesized that this new neoadjuvant chemotherapy followed by surgery and chemoradiation therapy would be well tolerated and would have a high curative resection rate.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary objective: To evaluate the tolerability and toxicity of neoadjuvant cisplatin plus paclitaxel and postoperative chemoradiation therapy with fluorouracil plus leucovorin calcium in patients with high-risk gastric cancer.

Secondary objectives: To assess the pathologic response of gastric tumors to neoadjuvant cisplatin plus paclitaxel chemotherapy, and preliminarily assess the patterns of failure and disease free and overall survival.

OUTLINE: Patients receive 3 courses of preoperative neoadjuvant chemotherapy given on day 1 every 21 days. Courses consist of an intravenous infusion of cisplatin and a 3 hour intravenous infusion of paclitaxel on day 1. Patients then undergo surgery for tumor removal on day 63, followed 4-6 weeks later by one course of daily intravenous bolus leucovorin calcium and fluorouracil for 5 days. Chemotherapy is repeated 4-6 weeks later for the first 4 days of week 1 and the last 3 days of week 5 of radiation therapy given 5 days a week for 5 weeks. Patients receive two more courses, 4 weeks apart, of fluorouracil and leucovorin calcium for 5 days 4-6 weeks after completing radiation treatment. Patients are followed every month for the first 3 months, every 3 months for the next 21 months, every 6 months for the next year, and annually thereafter.

PROJECTED ACCRUAL: Approximately 30-42 patients will be accrued over 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction
* Localized cancer that is potentially curable by surgery (T2, N1-2, M0 or T3-4, any N, M0)
* No metastatic cancer to the ovaries
* Age: 18 and over
* Easter Cooperative Oncology Group (ECOG) performance status 0-2
* White blood cell (WBC) count at least 4,000 cells/mm3
* Platelet count at least 150,000/mm3
* Bilirubin less than 2 mg/dL
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance greater than 50 mL/min
* Caloric intake must be at least 1500 kcal/day
* No prior history of cancer within the past 5 years except for basal cell carcinoma of the skin or in situ carcinoma of the cervix
* No prior radiation therapy, except for skin cancer
* Fertile patients must use adequate contraception
* Met criteria for re-registration after surgery

  * T1N1-2M0, T2N1-2M0 or T3-4NanyM0 at time of initial re-registration.
  * No evidence of metastatic disease from postoperative pathologic staging.
  * ECOG performance status of 0, 1, or 2 at re-registration
  * Curative resection performed
  * Re-registered 4 - 6 weeks from the date of surgery
  * WBC ≥ 4000 cells/mm³, platelets ≥ 150,000/mm³, creatinine ≤ 1.5 mg/dl or creatinine clearance of > 50 ml/min (measured or calculated) and total serum bilirubin < 2 mg/dl, all within four weeks prior to re-registration

Exclusion Criteria:

* Prior chemotherapy
* Clinically significant auditory impairment
* Significant heart disease
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1999-06-01 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David I. Rosenthal, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (30):
- United States (30):
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - New England Medical Center Hospital, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin

REFERENCES:
- [Result] Chakravarthy AB, Catalano PJ, Mondschein JK, Rosenthal DI, Haller DG, Whittington R, Spitz FR, Wagner H, Sigurdson ER, Tschetter LK, Bayer GK, Mulcahy MF, Benson AB. Phase II Trial of Paclitaxel/Cisplatin Followed by Surgery and Adjuvant Radiation Therapy and 5-Fluorouracil/Leucovorin for Gastric Cancer (ECOG E7296). Gastrointest Cancer Res. 2012 Nov;5(6):191-7. PMID 23293700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E7296 was activated on February 25, 1999, accrued its first patient on June 1, 1999, and terminated on March 18, 2002 with a final accrual of 39 patients (accrual goal: 42 patients) enrolled by 13 ECOG affiliated institutions.
Groups:
- Experimental Arm: Patients receive 3 courses of preoperative neoadjuvant chemotherapy (an intravenous infusion of cisplatin and a 3 hour intravenous infusion of paclitaxel) given on day 1 every 21 days. Patients then undergo surgery for tumor removal on day 63, followed 4-6 weeks later by one course of daily intravenous bolus leucovorin calcium and fluorouracil for 5 days. Chemotherapy is repeated 4-6 weeks later for the first 4 days of week 1 and the last 3 days of week 5 of radiation therapy given 5 days a week for 5 weeks. Patients receive two more courses, 4 weeks apart, of fluorouracil and leucovorin calcium for 5 days 4-6 weeks after completing radiation treatment.
Period: Step 1 (Neoadjuvant Therapy)
Arm/Group | Experimental Arm
Started | 39
Eligible and Treated | 38
Complete 3 Cycles of Neoadjuvant Therapy | 35
Completed | 35
Not Completed | 4
Not completed — Ineligible for step 1 | 1
Not completed — Adverse Event | 3
Period: Surgery
Arm/Group | Experimental Arm
Started | 35
Completed | 28 (1 patient did not complete neoadjuvant therapy but went to surgery anyway, not included here.)
Not Completed | 7
Not completed — Unresectable at surgery | 3
Not completed — Progression before surgery | 2
Not completed — Unevaluable and off study | 2
Period: Re-register to Step 2 After Surgery
Arm/Group | Experimental Arm
Started | 28
Completed | 10
Not Completed | 18
Not completed — Less than 15 nodes examined | 7
Not completed — Positive margins | 5
Not completed — Other complications | 2
Not completed — Reason unknown | 1
Not completed — Ineligible due to tumor staging | 3
Period: Step 2 (Adjuvant Therapy)
Arm/Group | Experimental Arm
Started | 10
Eligible and Treated on Step 2 | 7
Completed | 4
Not Completed | 6
Not completed — Ineligible | 1
Not completed — Death | 1
Not completed — Progression before starting treatment | 1
Not completed — Excessive complication | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated in step 1
Arm/Group | Experimental Arm
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 57 [34 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Secondary Outcome: Best Confirmed Response to Neoadjuvant Therapy
Description: Response was based on pathology at surgery. A patient achieved complete response if no gross or microscopic tumor were identified with the surgical specimen and nodal tissue. Stable response was defined as a response that did not qualify as complete response or progressive disease (PD), where PD indicated metastatic spread. Best confirmed response rate was defined as the proportion of patients with complete response (CR). A patient was considered unevaluable if the patient did not have surgery, the pathologist did not examine at least 15 lymph nodes, or the pathology report was unavailable.
Time Frame: Assessed at surgery time (surgery performed during week 8-10 after registration to the study)
Population: Eligible and treated patients on step 1. Since no patient had a complete response in the study, one-sided 95% confidence interval was provided here.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 38
percentage of participants | 0 [0 to 7.58]

2. Primary Outcome: Grade 3 or Higher Toxicity Incidence on Step 1
Description: Incidence is defined as proportion of patients with any grade 3 or higher treatment-related toxicities among all treated patients.
Time Frame: assessed at the end of every cycle (cycle=21 days) during treatment (3 cycles in total)
Population: eligible and treated patients on step 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 38
percentage of participants | 65.8 [48.6 to 80.4]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from registration to death, where a subject was censored on date of last record alive.
Time Frame: assessed every month for the first 3 months, every 3 months for the next 21 months, every 6 months for the next year, and annually thereafter up to year 10
Population: eligible and treated patients on step 1
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Experimental Arm
Number analyzed (Participants) | 38
years | 1.55 [1.24 to 2.23]

4. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) was defined as time from registration until progression, recurrence, or death, whichever occurred first. If date of death occurred beyond three months from the date of last disease assessment, then PFS was censored at date of last disease assessment. Patients who were alive and progression-free were censored at the date of last disease evaluation.
Time Frame: as for outcome 3
Population: eligible and treated patients on step 1
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Experimental Arm
Number analyzed (Participants) | 38
years | 0.68 [0.35 to 1.43]

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment and for 30 days after the end of treatment
Groups:
- Step 1(Neoadjuvant Therapy): Patients receive 3 courses of preoperative neoadjuvant chemotherapy given on day 1 every 21 days. Courses consist of an intravenous infusion of cisplatin and a 3 hour intravenous infusion of paclitaxel on day 1.
- Step 2 (Adjuvant Therapy): After neoadjuvant therapy, patients undergo surgery for tumor removal on day 63, followed 4-6 weeks later by one course of daily intravenous bolus leucovorin calcium and fluorouracil for 5 days. Chemotherapy is repeated 4-6 weeks later for the first 4 days of week 1 and the last 3 days of week 5 of radiation therapy given 5 days a week for 5 weeks. Patients receive two more courses, 4 weeks apart, of fluorouracil and leucovorin calcium for 5 days 4-6 weeks after completing radiation treatment.
Arm/Group | Step 1(Neoadjuvant Therapy) | Step 2 (Adjuvant Therapy)
Serious Adverse Events (participants affected / at risk) | 25/38 | 6/7
Other Adverse Events (participants affected / at risk) | 38/38 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1(Neoadjuvant Therapy) (N=38) | Step 2 (Adjuvant Therapy) (N=7)
Anaphylaxis (Immune system disorders) | 1 | 0
White blood cell decreased (Investigations) | 4 | 3
Neutrophil count decreased (Investigations) | 18 | 5
Platelet count decreased (Investigations) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Weight loss (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 2
Alkaline phosphatase increased (Investigations) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Creatinine increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1(Neoadjuvant Therapy) (N=38) | Step 2 (Adjuvant Therapy) (N=7)
Hearing impaired (Ear and labyrinth disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 2
White blood cell decreased (Investigations) | 29 | 7
Neutrophil count decreased (Investigations) | 16 | 5
Platelet count decreased (Investigations) | 9 | 4
Cardiac disorders - Other (Cardiac disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1
Fatigue (General disorders) | 28 | 5
Fever (General disorders) | 2 | 0
Weight loss (Investigations) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 4
Nail loss (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 13 | 2
Constipation (Gastrointestinal disorders) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 29 | 6
Mucositis oral (Gastrointestinal disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 20 | 2
Diarrhea (Gastrointestinal disorders) | 16 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 | 0
Alkaline phosphatase increased (Investigations) | 5 | 2
Blood bilirubin increased (Investigations) | 3 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 6 | 1
Anxiety (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 13 | 0
Watering eyes (Eye disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 0
Pain (General disorders) | 2 | 1
Creatinine increased (Investigations) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less